CLINICAL TRIAL: NCT01848301
Title: Endothelial Injury and Development of Coronary Intimal Thickening After Heart Transplantation
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: loss of funding
Sponsor: Gladwin, Mark, MD (Individual)
Responsible Party: Principal Investigator, Catalin Toma, MD, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO12060201; American Heart Association (Other Grant/Funding Number: 12CRP11550009)
Record Dates: First submitted 2013-05-02; First posted 2013-05-07 (Estimated); Last update posted 2017-09-06 (Actual); Status verified 2017-09

CONDITIONS: Cardiac Allograft Vasculopathy; Antibody Mediated Rejection
Keywords: Optical Coherence Tomography; OCT; Coronary Allograft Vasculopathy; Donor Specific Antibodies; Acetylcholine; Coronary endothelial function; Brachial Artery Flow Mediated Dilation; Heart transplantation
MeSH Terms: interventions — Tomography, Optical Coherence; Acetylcholine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single arm (Experimental): All subjects will undergo a Brachial Artery Flow Medicated Dilation prior to heart catheterization. After routine heart catheterization, images of their coronary artery will be recorded by Optical Coherence Tomography (OCT) during infusion of Acetylcholine.
  Interventions: Device: Optical Coherence Tomography; Drug: Acetylcholine; Procedure: Brachial Artery Flow Mediated Dilation

INTERVENTIONS:
Device: Optical Coherence Tomography — OCT imaging of the LAD coronary artery
  Other Names: OCT
Drug: Acetylcholine — Infusion in the coronary artery to study endothelial function
  Other Names: Miochol; Miochol-e
Procedure: Brachial Artery Flow Mediated Dilation — Assess peripheral brachial artery endothelial function

SUMMARY:
Coronary allograft vasculopathy (CAV) is the leading cause of late graft failure and second leading cause of late mortality after heart transplantation. CAV has been associated with a variety of traditional risk factors for atherosclerosis; however, immune mediated injury from development of de-novo donor-specific antibodies after transplantation also likely plays an important role. Similar to the progression of traditional atherosclerosis, it is likely that endothelial dysfunction is the precursor to the development of intimal thickening and CAV.

The investigators hypothesize that coronary allograft vasculopathy after heart transplantation as defined by progressive neointimal hyperplasia is preceded by endothelial dysfunction, which in turn is at least partly mediated by donor specific antibodies.

The investigators are proposing a prospective study in humans to test the above hypothesis and further mechanistically understand how CAV progresses. In this study the investigators will test for coronary endothelial function by infusing acetylcholine into the coronary artery and measure intimal hyperplasia by optical coherence tomography (OCT) and compare findings in patients with and without donor specific antibodies.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 1 year post heart transplantation
* Subjects will include both male and females
* Be at least 18 years of age

Exclusion Criteria:

* Known coronary artery disease after transplantation
* Evidence of strong or moderate antibodies already present at the time of the transplant
* Severe renal dysfunction defined as creatinine clearance of <30 or on hemodialysis.
* 3 or more episodes of acute cellular rejection
* Females who are pregnant
* Patients requiring endomyocardial biopsy at the time of catheterization
* Patients unable to tolerate heparin or systemic anticoagulation
* History of multi-organ transplant
* Patients unable to give consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-09; Primary Completion 2014-09 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be a comparison of intimal thickness in the coronary artery by Optical Coherence Tomography with presence or absence of donor specific antibodies. | baseline (year 1 post transplant) and annually for 2 years

SECONDARY OUTCOMES:
Assessment of epicardial coronary endothelial function by measuring change in vessel size in response to acetylcholine and how this compares to peripheral endothelial function. | baseline (year 1 post transplant) and annually for 2 years
Prospectively determine the association of HLA and non-HLA donor specific antibodies that activate complement with endothelial dysfunction and intimal thickening. | baseline (year 1 post transplant) and annually for 2 years
Gene expression of white blood cells by microRNA and how this relates to endothelial function and intimal thickness. | baseline (year 1 post transplant) and annually for 2 years
Plaque characterization in coronary artery by OCT | baseline (year 1 post transplant) and annually for 2 years
Natural progression of coronary allograft vasculopathy over first 2 years after transplantation | baseline (year 1 post transplant) and annually for 2 years
Comparison of endothelial function in the coronary artery with presence or absence of donor specific antibodies. | baseline (year 1 post transplant) and annually for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Catalin Toma, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Khandhar SJ, Yamamoto H, Teuteberg JJ, Shullo MA, Bezerra HG, Costa MA, Selzer F, Lee JS, Marroquin OC, McNamara DM, Mulukutla SR, Toma C. Optical coherence tomography for characterization of cardiac allograft vasculopathy after heart transplantation (OCTCAV study). J Heart Lung Transplant. 2013 Jun;32(6):596-602. doi: 10.1016/j.healun.2013.02.005. Epub 2013 Mar 15. PMID 23499356